CLINICAL TRIAL: NCT04690478
Title: Remote Blood Pressure Management Clinical Application Research
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: The Affiliated Hospital of Qingdao University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 20-3-4-54-nsh
Record Dates: First submitted 2020-12-08; First posted 2020-12-30 (Actual); Last update posted 2022-02-17 (Actual); Status verified 2022-02

CONDITIONS: Hypertension
Keywords: Hypertension;; Telemedicine;; Remote blood pressure monitoring
MeSH Terms: conditions — Hypertension

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Remote blood pressure management group (Experimental): Remote blood pressure management group through remote blood pressure management the platform realizes functions such as automatic upload of patient measurement data, intelligent analysis, and early warning reminders
  Interventions: Device: Electronic remote blood pressure monitor
- Non-remote blood pressure management group (Other): Non-remote blood pressure management group is distributed a set of ordinary household electronic sphygmomanometer, and the blood pressure is recorded by themselves at home following routine community office follow-up
  Interventions: Device: Ordinary household electronic sphygmomanometer
- Routine blood pressure management group (Other): Routine blood pressure management group follows routine community office follow-up and uses office electronic sphygmomanometer to measure blood pressure
  Interventions: Device: Office electronic sphygmomanometer

INTERVENTIONS:
Device: Electronic remote blood pressure monitor — Remote blood pressure management group through remote blood pressure management the platform realizes functions such as automatic upload of patient measurement data, intelligent analysis, and early warning reminders
  Arms: Remote blood pressure management group
Device: Ordinary household electronic sphygmomanometer — One group is distributed a set of ordinary household electronic sphygmomanometer, and the blood pressure is recorded by themselves at home following routine community office follow-up
  Arms: Non-remote blood pressure management group
Device: Office electronic sphygmomanometer — One group follows routine community office follow-up and uses office electronic sphygmomanometer to measure blood pressure
  Arms: Routine blood pressure management group

SUMMARY:
Recruit patients with essential hypertension and randomly divide them into three groups. For 24 months, observe the patient's blood pressure level and blood pressure compliance rate,Risk assessment, etc.

DETAILED DESCRIPTION:
Recruit patients with essential hypertension and randomly divide them into three groups. One group through remote blood pressure management platform realizes functions such as automatic upload of patient measurement data, intelligent analysis, and early warning reminders;One group is distributed a set of electronic sphygmomanometers , and the blood pressure is recorded by themselves following routine community hypertension management; one group follows routine community hypertension management. For 24 months, observe the patient's blood pressure level and blood pressure compliance rate,Risk assessment, etc. The main technical difficulties and problems to be solved: Widely popularize remote blood pressure based on "Cloud Sharing Smart Cabinet" Management mode. Innovation point: Provide primary hospitals with an intelligent, simple and efficient innovative tool for the management of residents chronic diseases, and improve the management level of chronic diseases in my country promotly; adopt intelligent terminal equipment to realize automatic data collection and transmission to ensure patient real blood pressure data timely and continuously, providing data reference and basis for academic research and the prevention and treatment of chronic diseases, and promoting scientific research in the prevention and treatment of chronic diseases in my country.

ELIGIBILITY:
Inclusion Criteria:

* Clinical diagnosis of primary hypertension
* Must be aged at ≥18 years old and ≤75 years old
* Must have a smart phone and have the ability to use smart devices
* Must be local permanent resident population who volunteered to participate in the study and received a 2-year follow-up
* Must sign informed consent

Exclusion Criteria:

* Participated in other clinical trials within 4 weeks before the start of this study
* The systolic blood pressure in the office was ≥180 mmHg, and/or the diastolic blood pressure was ≥110 mmHg
* Uremia, creatinine>250umol/l
* History of acute heart disease in the past three months
* Terminal diseases such as malignant tumors
* Severe cognitive impairment
* Severe diabetes patients (glycated hemoglobin>11%)
* Severe valvular heart disease, cardiomyopathy, and poor heart function
* Atrial fibrillation and atrioventricular block
* Arm circumference >35cm or <26cm
* Spouse or relatives have been included in this research
* Pregnant or breastfeeding women
* Live in an unfixed state

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 1050 (Estimated)
Dates: Start 2020-06-01 (Actual); Primary Completion 2023-03-31 (Estimated); Study Completion 2023-06-30 (Estimated)

PRIMARY OUTCOMES:
Blood pressure level(SBP and DBP) | 2years
  Blood pressure level(SBP and DBP)
Blood pressure compliance rate(SBP and DBP) | 2years
  Blood pressure compliance rate(SBP and DBP)
Cardiovascular risk assessment | 2years
  Cardiovascular risk assessment
Economic benefit | 2years
  Compare economic benefit among the three groups by counting the cost of hypertension treatment and the cost of hospitalization due to complications of hypertension of patients in every group.
improved level of quality of life | 2years
  Compare improved level of quality of life among the three groups by counting the proportions of patients with improvement of lifestyle and living habits in every group.The content of improvement of lifestyle and living habits mainly including reduction of the frequency and amount of smoking, drinking, high-salt diet and high-fat diet, increase of the frequency and amount of exercise, and so on.
Clinical prognosis assessment | 2years
  Compare clinical prognosis among the three groups by counting incidence of non-fatal acute myocardial infarction, non-fatal stroke, hospitalization for unstable angina, hospitalization for worsening heart failure in every group.
Therapeutic compliance | 2years
  Compare therapeutic compliance among the three groups by counting the proportions of patients taking medication on time and regularly receiving follow-up at office in every group.

CONTACTS AND LOCATIONS:
Overall Officials: Yu haichu, master, Study Chair — Affiliated Cardiovascular Hospital of Qingdao University
Locations (1):
- Remote electronic sphygmomanometer, Qingdao, Shandong, China

REFERENCES:
- [Derived] Teng TQ, Sun GX, Yu ZY, Liu ZS, Wang T, Wu Q, Qin RR, Wang MM, Chen R, Xu JC, Zhang N, Song BX, Liu X, Zhang YY, Yu HC. Efficiency of remote monitoring and guidance in blood pressure management: a randomized controlled trial : The role of remote monitoring in improving hypertension management. BMC Med. 2025 Aug 5;23(1):459. doi: 10.1186/s12916-025-04278-6. PMID 40764960

DOCUMENTS (2):
  • Study Protocol (2020-05-01): https://cdn.clinicaltrials.gov/large-docs/78/NCT04690478/Prot_000.pdf
  • Informed Consent Form (2020-05-01): https://cdn.clinicaltrials.gov/large-docs/78/NCT04690478/ICF_001.pdf